CLINICAL TRIAL: NCT04467723
Title: CAFs (Combination of Atezolizumab and Pirfenidone in Second-line and Beyond NSCLC): a Phase I/II Study
Brief Title: Combination of Atezolizumab and Pirfenidone in Second-line and Beyond NSCLC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: parkview cancer institute (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2020-CAFs
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: NSCLC Stage IV; NSCLC, Recurrent
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Recurrence | interventions — atezolizumab; pirfenidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Atezolizumab (Tecentriq) intravenous (IV) 1200mg flat dose day 1 then every 3 weeks.
  Pirfenidone (Esbriet) orally (PO) with food according to this schedule:
  Days 1-14: 267 milligrams (mg) orally three times per day (PO TID) Days 15-29: 534 mg PO TID Days 30 onward until progression: 801 mg PO TID
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab is given as an intravenous infusion at 1200 mg every 3 weeks. Pirfenidone is taken by mouth 3 times a day with the dose increasing every 2 week until day 30
  Other Names: Pirfenidone

SUMMARY:
The purpose of this study is to see if adding pirfenidone to atezolizumab will increase anti tumor activity and reduce treatment resistance in stage 4 and recurrent non- small cell lung cancer participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant or legal representative is able to provide written informed prior to performing any protocol-related procedures
* Is willing and able to comply with scheduled visits, treatment schedule, laboratory testing and other requirements of the study
* Men or women at least 18 years of age with histologically or cytologically confirmed non-small cell lung cancer
* Previous history of other than lung cancer is allowed if no active treatment for that cancer within 1 year
* Life expectancy of at least 6 months
* De novo stage IV or recurrent NSCLC without actionable mutation (e.g. EGFR/ ALK/ ROS-1) that was previously treated with either PD-1 / PD-L1 or the combination of PD1/PDL1 and cytotoxic chemotherapy, no more than 2 systemic regimens for metastatic disease with measurable disease *. Maintenance therapy will be considered part of the 1 regimen
* At least 1 measurable lesion
* PDL1 TPS score less than 1% or unknown: first-line must be PD1/PDL1 inhibitor in combination with chemotherapy
* Early stage (I-III) NSCLC treated with adjuvant or neoadjuvant chemotherapy then PD1/PDL1 inhibitor treatment for recurrent disease
* Recurrent Unresectable stage III NSCLC treated with prior chemoradiation followed by maintenance PD1/PDL1 inhibitor with measurable disease
* Eastern Cooperative Group (ECOG) Performance Status 0 - 2
* Is able to swallow oral medications
* Adequate hematologic function
* Adequate organ function

Exclusion Criteria:

* The presence of any other concurrent severe and/or uncontrolled medical condition that would, in the investigator or treating physician's judgement, cause unacceptable safety risks, contraindicate patient participation in the clinical study or compromise compliance with the protocol
* Has received investigational agents within 14 days or 5 half-lives of the compound or active metabolites, whichever is longer, before the first dose of study treatment
* Has a known hypersensitivity to atezolizumab or pirfenidone
* Has active medical or psychiatric illness that would interfere with the study treatment
* Has uncontrolled diabetes
* Has any of the following cardiac diagnoses:

Unstable angina Myocardial infarction within 6 months Uncontrolled congestive heart failure Left ventricular ejection fraction < 35%

* Has a history of any Grade 3 or 4 toxicities to a prior checkpoint inhibitor treatment
* Is pregnant or breast feeding
* Uncontrolled HIV
* Clinically diagnosed with grade 2 or 3 radiation-induced lung injury within the last 3 months prior to registering for the study
* Has a history of idiopathic pneumonitis that required systemic agent including steroid
* Has drug-induced pneumonitis
* Has evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Smoker of more than 1 pack / day
* Has active peptic ulcer diagnosed within 4 weeks of enrollment
* Active infection requiring systemic treatment
* Current use of systemic antibacterial or antifungal agent
* Prior monoclonal antibody within 4 weeks before study Day 1 Exception: The use of denosumab
* Patient not recovered to ≤ Grade 1 from AEs due to agents administered more than 4 weeks earlier
* Concurrent use of other investigational agents
* Uncontrolled or symptomatic brain metastasis or leptomeningeal disease that requires use of steroids
* Use of strong CYP1A2 inhibitors
* Previous history of cancer with active treatment within less than 1 year of enrollment
* Active auto-immune diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Grade 3 toxicity | Cycle 1 day 1 to Cycle 3 day 1 (Each cycle is 21 days)
  CTCAE v5.0
Occurrence of Grade 4 toxicity | Cycle 1 day 1 to Cycle 3 day 1 (Each cycle is 21 days)
  CTCAE v5.0

SECONDARY OUTCOMES:
Overall response rate (ORR) of participants | Cycle 1 day 1 to Cycle 3 day 1 (Each cycle is 21 days)
  RECIST 1.1
Progression Free Survival (PFS) | From Cycle 1 day 1 (Each cycle is 21 days) for up to 2 years after end of treatment
  RECIST 1.1
1-year overall survival (OS) rate: Proportion of participants alive at 1 year from Cycle 1 day 1 | Cycle 1 day 1 up to 1 year post-Cycle 1 day 1 (Each cycle is 21 days)
  Medical records

CONTACTS AND LOCATIONS:
Overall Officials: Chao Huang, MD, Principal Investigator — The University of Kansas
Locations (2):
- United States (2):
  - The University of Kansas Cancer Center (KUCC), Fairway, Kansas
  - The University of Kansas Cancer Center, Westwood Campus, Kansas City, Kansas

IPD SHARING:
Plan to Share IPD: No